CLINICAL TRIAL: NCT03382184
Title: Fractional Photothermolysis for the Treatment of Hair Loss
Brief Title: Fractional Photothermolysis for Hair Follicle Induction
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Natasha Mesinkovska, Principal Investigator, University of California, Irvine
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20173385
Record Dates: First submitted 2017-12-13; First posted 2017-12-22 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Alopecia
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Intervention Model Description: This is a prospective, dual-arm study involving the Fraxel DUAL or Halo laser for the regrowth of hair after alopecia.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Fraxel DUAL 1550 nm (Experimental): The Fraxel DUAL 1550 nm laser will be used at 7 mJ, 8 pulses, 120 spots/cm2, treatment level 3 (9% coverage) for hair regrowth. 25 patients with alopecia will be part of this group.
  Interventions: Device: Fraxel Dual laser
- Halo Hybrid Laser 1550 nm (Experimental): The Halo laser will be used per protocol due to the dynamic thermal optimization technology for hair regrowth. 25 patients with alopecia will be part of this group.
  Interventions: Device: Halo laser

INTERVENTIONS:
Device: Fraxel Dual laser — The Fraxel DUAL 1550 nm laser will be used at 7 mJ, 8 pulses, 120 spots/cm2, treatment level 3 (9% coverage) for hair regrowth.
  Arms: Fraxel DUAL 1550 nm
Device: Halo laser — The Halo hybrid laser will be used per protocol due to its dynamic thermal optimization technology for hair regrowth.
  Arms: Halo Hybrid Laser 1550 nm

SUMMARY:
This study is being done to evaluate the effects of fractional photothermolysis (known as laser resurfacing) using fractional laser for the induction of hair follicles via skin rejuvenation in subjects with scalp alopecia (specifically, alopecia on the superior forehead at the frontal hairline). Fractional photothermolysis has been shown to be effective in promoting hair growth. The investigators will study 50 subjects who will be treated 6-10 times at 2-4 week intervals. Each participant will have half of their head treated with a laser, either Fraxel DUAL 1550 or Halo by Sciton, and the other half of their head will be left untreated as a control. Half of the individuals will randomly be assigned to the group to be treated with Fraxel DUAL 1550, and the other half will be treated with Halo by Sciton. Visual observation and digital, photographic, non-invasive imaging will be used to compare the treated and untreated area to assess for differences in hair follicle stimulation rates, number and density of hairs.

As noted above, the types of lasers we plan to use include the non-ablative fractional laser settings for the Fraxel DUAL 1550 and Halo by Sciton. A fractional laser is a laser that directs an intense burst of laser energy on the skin. The treatment deposits heat deep into the dermis to tighten skin and stimulate collagen remodeling. The necrotic (death of cells or tissue) injury heals rapidly and adverse effects are few. Laser resurfacing is commonly used for rejuvenation of the skin to improve quality, tone, and texture.

DETAILED DESCRIPTION:
Introduction Alopecia is also known as hair loss, and it occurs due to aging, nutritional or hormonal imbalance, or immune system etiology. It affects both males and females of different ages and races. Hair may fall out in clumps, break off leaving short stubs, or become thinner over time. The alopecia can be of a scarring or non-scarring nature. The most common form of hair loss is non-scarring, or noncicatricial, alopecia. In this case, the damage is not permanent, and although hair loss cannot be cured, it can be treated. Hair loss is usually not a sign of an underlying medical disorder. However, hair loss may affect self-esteem and cause anxiety affecting the quality of life. Scarring, or cicatricial, alopecia is a rare disorder that destroys the hair follicle and replaces it with scar tissue, resulting in permanent hair loss.

Causes

There are many genes that contribute to hair loss, so it can be hereditary. There are also other causes, including:

* Thyroid disorders
* Pregnancy
* Anemia
* Autoimmune diseases like polycystic ovarian syndrome
* Skin conditions like Psoriasis and seborrheic dermatitis

Treatment Options Topical Minoxidil (Rogaine) and anti-inflammatory medications, such as topical and intra-lesional steroids, are used for alopecia. It is a solution that is applied directly to the scalp to stimulate the hair follicle. It slows hair loss, and some people grow new hair. Hair loss returns when the medication is stopped.

Finasteride is a prescription medicine that interferes with the production of a highly active form of testosterone that is linked to baldness. It slows hair loss. It works slightly better than minoxidil. Hair loss returns when you stop using the medicine. This prescription medication is also sometimes given to women who have been through menopause. Its role in female pattern hair loss is controversial, with both success and failure reported to occur.

Dutasteride is similar to finasteride, but may be more effective.

Hair transplants are also an option, though they are invasive and expensive. It consists of removing tiny plugs of hair from areas where the hair is continuing to grow and placing them in areas that are balding. This can cause minor scarring and possibly infection.

New Therapy Fractional photothermolysis was originally designed as a form of laser therapy to treat wrinkles and scars. Although the link between laser treatment and hair growth is not clear and the exact mechanism still unknown, there is evidence to support that laser irradiation holds potential for the induction of hair follicles in subjects with alopecia. Laser therapy has been reported to increase hair growth and activate hair follicles. The lasers rejuvenate skin, and hair follicles are a part of skin, along with nails, so through the rejuvenation of skin, these things also get rejuvenated. Clinical examples of photo-induced hair growth include the paradoxical hair growth after laser hair removal, and hair growth after some level of wound healing by lasers has been performed. Several studies have been performed, analyzing the effectiveness of laser treatment of different settings, and researchers have observed an increase in hair numbers and density on the treatment side of the head. Improvements were most notable when the laser settings followed a low energy and high density protocol. A review of the literature demonstrates that more research needs to be done on this topic, but fractional photothermolysis may be a new, effective way to treat different types of hair loss. The types of lasers the investigators plan to use include Fraxel restore and Sciton Halo, a fractional hybrid laser that combines fractional erbium ablative lasers with a fractional non-ablative laser. The use of the fractional photothermolysis Fraxel laser and Sciton Halo laser have been approved by the FDA for treatment of the hands, face, and body. Fraxel received aesthetic clearance in November 2003.

These lasers do not meet the definition of a significant risk device because the investigators do not believe that they present a potential for serious risk to the health, safety, or welfare of a subject. Side effects that have been reported from use with these lasers include redness and tenderness in the area that it was applied, and these side effects don't last more than a couple days. These lasers do not impair human health.

ELIGIBILITY:
Inclusion Criteria:

* Must be between the ages of 18 to 90 years old
* Diagnosed with hair loss on scalp by a dermatology
* No other treatments for hair loss have been done in the past 1 month
* No evidence of spontaneous hair growth
* Good health
* Must agree to comply with study treatment and protocol
* Healthy scalp without evidence of neoplasm
* Scarring and/or non-scarring alopecia acceptable

Exclusion Criteria:

* Any visible signs of neoplasm, infection, inflammatory disease of the scalp
* No history of photosensitivity, impaired wound healing, chronic liver or kidney disease
* No concurrent use of minoxidil/Rogaine, platelet-rich plasma (PRP), or light devices for hair regrowth
* Has not initiated use of finasteride/Propecia or spironolactone in the 3 months preceding the study

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-10-20 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Hair regrowth by dermoscopy | 24 weeks
  Hair will be counted before and after treatment using dermoscopy on both the treated and untreated scalp.
Hair regrowth by optical coherence tomography (OCT). | 24 weeks
  Hair will be counted before and after treatment using OCT on both the treated and untreated scalp.

SECONDARY OUTCOMES:
Hair regrowth impact on Quality of Life | 24 weeks
  Patients will be asked how hair regrowth has affected their quality of life over the period of 12 weeks of treatment and then 12 weeks of follow-up using a Likert scale (0-10).

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, Irvine, Department of Dermatology, Dermatology Clinical Research Center, Hewitt Hall, Irvine, California, United States

IPD SHARING:
Plan to Share IPD: No
Currently there is no plan to share individual participant data with other researchers.

REFERENCES:
- [Background] Kim WS, Lee HI, Lee JW, Lim YY, Lee SJ, Kim BJ, Kim MN, Song KY, Park WS. Fractional photothermolysis laser treatment of male pattern hair loss. Dermatol Surg. 2011 Jan;37(1):41-51. doi: 10.1111/j.1524-4725.2010.01833.x. Epub 2010 Dec 28. PMID 21199096
- [Background] Lee GY, Lee SJ, Kim WS. The effect of a 1550 nm fractional erbium-glass laser in female pattern hair loss. J Eur Acad Dermatol Venereol. 2011 Dec;25(12):1450-4. doi: 10.1111/j.1468-3083.2011.04183.x. Epub 2011 Aug 4. PMID 21812832
- [Background] Bae JM, Jung HM, Goo B, Park YM. Hair regrowth through wound healing process after ablative fractional laser treatment in a murine model. Lasers Surg Med. 2015 Jul;47(5):433-40. doi: 10.1002/lsm.22358. Epub 2015 May 6. PMID 25945952
- [Background] Update on fractional laser technology. J Clin Aesthet Dermatol. 2010 Jan;3(1):42-50. No abstract available. PMID 20725538
- [Background] Mlacker S, Aldahan AS, Simmons BJ, Shah V, McNamara CA, Samarkandy S, Nouri K. A review on laser and light-based therapies for alopecia areata. J Cosmet Laser Ther. 2017 Apr;19(2):93-99. doi: 10.1080/14764172.2016.1248440. Epub 2017 Jan 25. PMID 27802065
- [Background] Gupta AK, Carviel J, Abramovits W. Treating Alopecia Areata: Current Practices Versus New Directions. Am J Clin Dermatol. 2017 Feb;18(1):67-75. doi: 10.1007/s40257-016-0230-4. PMID 27770310